CLINICAL TRIAL: NCT06174922
Title: A Randomized Trial Comparing the Role of Prednisolone, Itraconazole, or Their Combination in Patients with Acute Stage of Allergic Bronchopulmonary Aspergillosis
Brief Title: A Randomized Trial of Prednisolone, Itraconazole, or Their Combination in Allergic Bronchopulmonary Aspergillosis
Acronym: PICA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Int/IEC/2023/SPL-1026A
Record Dates: First submitted 2023-11-24; First posted 2023-12-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Prednisolone; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prednisolone (Active Comparator): Oral prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper 5 mg every 4 weeks and discontinue by 4 months. After breakfast, oral prednisolone will be administered as a morning dose (8-10 am).
  Interventions: Drug: Prednisolone
- Itraconazole (Active Comparator): Oral SUBA-itraconazole 65 mg 2 capsules BD for 4 months. Oral itraconazole will be given twice daily (9 am and 9 pm) spaced one hour with meals. We will perform therapeutic drug monitoring for itraconazole at two weeks and two months. We will increase the itraconazole dose to a maximum of 390 mg/day (six 65 mg capsules) in those with trough itraconazole levels <0.5 µg/mL.
  Interventions: Drug: Itraconazole
- Prednisolone plus itraconazole (Experimental): Oral prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper 5 mg every 4 weeks and discontinue by 4 months. After breakfast, oral prednisolone will be administered as a morning dose (8-10 am); and, Oral SUBA-itraconazole 65 mg 2 capsules BD for 4 months. Oral itraconazole will be given twice daily (9 am and 9 pm) spaced one hour with meals. We will perform therapeutic drug monitoring for itraconazole at two weeks and two months. We will increase the itraconazole dose to a maximum of 390 mg/day (six 65 mg capsules) in those with trough itraconazole levels <0.5 µg/mL.
  Interventions: Drug: Prednisolone; Drug: Itraconazole

INTERVENTIONS:
Drug: Prednisolone — Prednisolone for 4 months
  Arms: Prednisolone; Prednisolone plus itraconazole
Drug: Itraconazole — SUBA-itraconazole for 4 months
  Arms: Itraconazole; Prednisolone plus itraconazole

SUMMARY:
The investigators hypothesize that a combination of prednisolone and itraconazole would significantly reduce the exacerbation rate at one-year of patients with acute allergic bronchopulmonary aspergillosis (ABPA) compared to itraconazole or prednisolone monotherapy.

In this study, 300 subjects aged ≥18 years with acute ABPA will be randomized to treatment with either prednisolone, itraconazole, or prednisolone plus itraconazole, all for four months each. After collecting baseline demographic, immunologic, and imaging data, the investigators will follow the patients every 2 months for the first two visits and then every four months for three visits. The primary outcome will be the proportion of subjects experiencing exacerbation (asthma or ABPA) 12 months after treatment completion.

DETAILED DESCRIPTION:
The principles of treating ABPA include using glucocorticoids to control the immunologic activity and antifungal agents to attenuate the fungal burden in the airways.4 Glucocorticoids are the first line treatment in acute stages of ABPA, although there are no placebo-controlled trials of glucocorticoids in ABPA. However, their effectiveness in ABPA is so well established that it might be considered unethical to conduct placebo-controlled trials. In one study, 92 subjects were randomized to receive high-dose (n=44) or low-dose (n=48) prednisolone. The numbers of subjects with exacerbation after one year (high-dose: 40.9% vs. medium-dose: 50%, p=0.59) were similar in the two groups. Although the composite response rates were significantly higher in the high-dose group, the improvement in lung function and the time to first exacerbation were similar in the two groups. [Eur Respir J. 2016;47(2):490-498] Specific antifungal agents in ABPA can modify the immune response by removing or reducing the antigenic stimulus consequent to a decreased fungal burden. Two randomized trials have recently shown that itraconazole and voriconazole monotherapies are as effective as prednisolone in treating acute-stage ABPA. [Chest. 2018;153(3):656-664|Eur Respir J. 2018;52(3):1801159] In the first randomized trial, 131 ABPA patients were randomized to receive either oral itraconazole (400 mg/day, [n=68]) or prednisolone (n=63) for four months. The proportion of subjects responding at six weeks was significantly higher in the prednisolone arm (100% vs. 88%; p=0.007). However, the number of subjects with exacerbations after one and two years of treatment was similar in the two groups. The time to first exacerbation was also similar in the two groups. The occurrence of adverse reactions was significantly higher in the glucocorticoid arm. Although prednisolone was more effective than itraconazole in inducing a response in acute-stage ABPA, itraconazole with fewer side effects is an acceptable alternative for treating acute-stage ABPA.[Chest. 2018;153(3):656-664] In the second trial, 50 ABPA patients were randomized to receive prednisolone (n=25) or voriconazole (n=25).[Eur Respir J. 2018;52(3):1801159] The response to treatment after six weeks and three months was similar in the two groups. The numbers of subjects with exacerbations after one year and two years were similar in the two groups. More recently, acute-stage ABPA subjects were randomized to receive either prednisolone (n=94) or prednisolone-itraconazole combination (n=97). The one-year exacerbation rate was 33% and 20.6% in the prednisolone and the prednisolone-itraconazole arms, respectively (p=0.054).[Eur Respir J. 2022;59(4):2101787] However, the study did not have a comparator arm of itraconazole monotherapy. Thus, it is unclear whether combination therapy is better than itraconazole or prednisolone monotherapy in reducing the occurrence of ABPA exacerbations.

The investigators hypothesize that the combination of prednisolone and itraconazole would significantly reduce the exacerbation rate at one-year than monotherapy. This study will compare the efficacy of prednisolone, itraconazole, or their combination in patients with acute stages of ABPA.

ELIGIBILITY:
Inclusion Criteria:

Consecutive subjects of acute stage allergic bronchopulmonary aspergillosis (ABPA) complicating asthma per the revised ISHAM-ABPA working group criteria

* newly diagnosed subjects with uncontrolled asthma or symptoms or radiology suggesting active lesions attributable to ABPA and meeting the diagnostic criteria of ABPA
* those previously meeting the diagnostic criteria for ABPA and presenting with sustained (≥2 weeks) clinical or radiological worsening; and increase in serum total IgE by ≥50% of the last recorded IgE value during clinical stability.

Exclusion Criteria:

* occurrence of ≥3 ABPA exacerbations in the last 18 months before enrollment
* contraindications to the use of either prednisolone or itraconazole
* subjects who have received oral prednisolone (or equivalent) ≥30 mg for ≥2 weeks or itraconazole (or voriconazole or posaconazole or isavuconazole) for more than 2 weeks, in the last 3 months
* chronic medical illnesses, including uncontrolled diabetes mellitus, chronic renal failure, chronic liver failure, chronic heart failure, and others
* patient on immunosuppressive drugs
* pregnancy
* enrollment in another trial of ABPA
* failure to provide informed consent
* asthma exacerbation: worsening respiratory symptoms for at least 24 hours without immunological or radiological deterioration of ABPA
* infective/bronchiectasis exacerbation: clinical deterioration for at least 24 hours with increase in cough; breathlessness; sputum volume or consistency; sputum purulence; fatigue, malaise, or fever; and hemoptysis without immunological or radiological deterioration of ABPA
* serologic ABPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Asthma or ABPA exacerbations | 12 months after treatment completion
  Proportion of subjects experiencing exacerbation (asthma or ABPA) 12 months after treatment completion

SECONDARY OUTCOMES:
Composite response | 8 weeks
  Proportion of subjects experiencing composite response defined as symptomatic improvement by at least 50%; and, major radiological improvement, and a decline in serum total IgE by at least 20% of baseline
IgE decline | 8 weeks
  Percentage decline in IgE (baseline IgE minus IgE after eight weeks/baseline IgE
Time to first ABPA exacerbation | 12 months after treatment completion
  Time to first ABPA exacerbation in days
Time to first asthma exacerbation | 12 months after treatment completion
  Time to first asthma exacerbation in days
Weight gain | Two months
  Treatment-related adverse effects
Hyperglycemia | Two months
  Treatment-related adverse effects
Cushingoid habitus | Two months
  Treatment-related adverse effects
Transaminitis | Two months
  Treatment-related adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Clinic, Dept. of Pulmonary Medicine, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided